CLINICAL TRIAL: NCT02702167
Title: The Dorsomedial Prefrontal Cortex as a Target in Treatment-resistant Bulimia Nervosa and Anorexia Nervosa: Investigating Target Engagement, Dosing, Reliability and Duration of Effect Using rTMS, fMRI, and a Sham Controlled Arm
Brief Title: High-frequency vs. Low-frequency vs. Sham DMPFC-rTMS for Bulimia and Anorexia Nervosa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic restrictions.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Blake Woodside, Psychiatrist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-6252-B
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Bulimia Nervosa; Anorexia Nervosa
Keywords: brain stimulation; rTMS
MeSH Terms: conditions — Bulimia Nervosa; Anorexia Nervosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-frequency rTMS (Experimental): 10 Hz repetitive transcranial magnetic stimulation to dorsomedial prefrontal cortex, once daily, 5 days per week for 6 weeks
  Interventions: Device: High-frequency rTMS
- Low-frequency rTMS (Experimental): 1 Hz repetitive transcranial magnetic stimulation to dorsomedial prefrontal cortex, once daily, 5 days per week for 6 weeks
  Interventions: Device: Low-frequency rTMS
- Sham rTMS (Sham Comparator): Sham repetitive transcranial magnetic stimulation to dorsomedial prefrontal cortex, once daily, 5 days per week for 6 weeks
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: High-frequency rTMS — 10 Hz active stimulation, once daily
  Other Names: Magventure Cool DB80 Active/Placebo Coil
  Arms: High-frequency rTMS
Device: Low-frequency rTMS — 1 Hz active stimulation, once daily
  Other Names: Magventure Cool DB80 Active/Placebo Coil
  Arms: Low-frequency rTMS
Device: Sham rTMS — Sham stimulation, once daily
  Other Names: Magventure Cool DB80 Active/Placebo Coil
  Arms: Sham rTMS

SUMMARY:
This trial will compare the efficacy and tolerability of 10 Hz vs. 1 Hz vs. sham repetitive transcranial magnetic stimulation targeting the dorsomedial prefrontal cortex, delivered once daily over 30 days, in patients with a diagnosis of bulimia or anorexia nervosa binge-purge subtype. The trial will include structural and functional MRI, and behavioral measures obtained before, during, and after treatment.

ELIGIBILITY:
Inclusion Criteria (Patient):

* Voluntary and Competent to Consent
* MINI confirmed Diagnosis of Bulimia Nervosa OR Anorexia Nervosa, Binge/Purge subtype
* Outpatient
* Between the ages of 18-65
* Have had no increase or initiation of any psychotropic medication in the last 4 weeks prior to screening
* Must adhere to research schedule.
* Pass the TMS Safety Screening Questionnaire.
* Failed to achieve a clinical response to at least one pharmacotherapy or behavioral treatment in the current episode.

Exclusion Criteria (Patient):

* Have a concomitant major unstable medical illness, cardiac pacemaker or implanted medical pump
* Have active suicidal intent
* Are pregnant
* Have a lifetime MINI diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform, delusional disorder, or current psychotic symptoms
* Have a MINI diagnosis of obsessive-compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia assessed by a study investigator to be primary and causing greater impairment than the ED
* Have received rTMS for any previous indication due to the potential compromise of subject blinding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Weekly Binge/Purge Frequency on Eating Disorder Examination (EDE) | Baseline, after each week of treatment, and 1, 4, 12, and 24 weeks post-treatment
  Outcome measured by a change in weekly binge and purge episodes from baseline to 2 weeks post-treatment. A 50% improvement in the score is considered a response to rTMS. A final score of 0 weekly binges and 0 weekly vomits is categorized as remission.

SECONDARY OUTCOMES:
Eating Disorder Inventory-3 | Baseline, after each week of treatment, and 1, 4, 12, and 24 weeks post-treatment
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline, after each week of treatment, and 1, 4, 12, and 24 weeks post-treatment

OTHER OUTCOMES:
Resting-state functional MRI | 1 week pre- and 1 week post-intervention
  10 min resting-state functional MRI acquisition at 3T

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Downar, MD PhD, Principal Investigator — University Health Network, Toronto; Blake Woodside, MD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided